CLINICAL TRIAL: NCT00665808
Title: Insulin Detemir (Levemir®) Versus Isophane (NPH) Insulin (Protaphane®) in Combination With Oral Antidiabetic Agents (OAD) in Patients With Diabetes Mellitus Type 2 Comparing Treatment Satisfaction, Diabetes-related and General Health-related Quality of Life, as Well as Diabetes-control
Brief Title: Observational Study on Treatment Satisfaction of Levemir® Versus Protaphane® During "Real-life" Usage in Germany
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1951
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: insulin detemir
- B
  Interventions: Drug: isophane human insulin

INTERVENTIONS:
Drug: insulin detemir — Observational study on treatment satisfaction of Levemir ® versus Protaphane® during "real-life" usage in Germany
  Other Names: Levemir®
  Groups: A
Drug: isophane human insulin — Observational study on treatment satisfaction of Levemir ® versus Protaphane® during "real-life" usage in Germany
  Groups: B

SUMMARY:
This NON INTERVENTIONAL OBSERVATIONAL STUDY is conducted in Europe. The purpose of this NON INTERVENTIONAL OBSERVATIONAL STUDY is to primarily investigate treatment satisfaction when using Levemir® versus Protaphane® in combination with OADs in daily settings.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from patient before first documentation of treatment in the observational study.
* Type 2 diabetes mellitus
* Patients, who should intensify treatment with long acting insulin in addition to their treatment with oral antidiabetic agents, due to insufficient blood glucose control
* No contraindication for use of Protaphane® or Levemir®

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients willing and able to give signed informed consent; Patients with Type 2 diabetes mellitus; Patients, who should intensify treatment with long acting insulin in addition to their treatment with oral antidiabetic agents, due to insufficient blood glucose control; Patients with no regular use of short acting insulin (occasional use for correction is allowed); Patients with no contraindication for use of Protaphane® or Levemir®
Sampling Method: Non-Probability Sample
Enrollment: 8125 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
treatment satisfaction (DTSQs and DTSQc) | over whole study duration, 24 weeks per patient

SECONDARY OUTCOMES:
diabetes-related quality of life (ADDQoL) | over whole study duration, 24 weeks per patient
general health-related quality of life (EQ-5D) | over whole study duration, 24 weeks per patient
Body weight | over whole study duration, 24 weeks per patient
metabolic control (HbA1c, fasting morning blood glucose) | over whole study duration, 24 weeks per patient
Insulin dose | over whole study duration, 24 weeks per patient
concomitant diabetes therapy (OADs) | over whole study duration, 24 weeks per patient
Hypoglycemia | over whole study duration, 24 weeks per patient
Adverse drug reactions, ADR | over whole study duration, 24 weeks per patient
Serious adverse drug reactions, SADR | over whole study duration, 24 weeks per patient
Pregnancy | over whole study duration, 24 weeks per patient

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mainz, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com